CLINICAL TRIAL: NCT00779818
Title: Electrical Acupuncture and Laser Therapy for Low Back Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Dr. John Zhang, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD1117060051
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Treatment by electrical acupuncture
  Interventions: Device: Electrical acupuncture
- Group 2 (Experimental): Treatment by laser
  Interventions: Device: Laser

INTERVENTIONS:
Device: Electrical acupuncture — Treatment by electrical acupuncture
  Arms: Group 1
Device: Laser — Treatment by laser
  Arms: Group 2

SUMMARY:
This is a treatment for low back pain using electrical stimulation and laser for 6 weeks.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effects of electroacupuncture and laser therapy to treat chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for over 6 weeks

Exclusion Criteria:

* Individuals with cancer
* Tuberculosis
* Pacemakers
* Pregnancy
* Osteoporosis
* Heart disease
* Kidney failure
* Thyroid disorders
* Diabetes
* Chronic disease
* Neurological diseases
* Skin or bleeding disorders
* Currently taking drugs or medications
* A health history questionnaire will be used to screen subjects

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Measure: Low Back Pain Disability Index, VAS Questionnaire, Revised Oswestry Pain Questionnaire | Before treatment and every two weeks for six weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States